CLINICAL TRIAL: NCT01959373
Title: Dysfunctions and Plasticity Mechanisms of Motor System Assessed by Cortico-cortical and Cortico-muscular Coherence Analysis in Amyotrophic Lateral Sclerosis
Status: Suspended | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-A00802-43; 2013-22 (Other: AP HM)
Record Dates: First submitted 2013-10-08; First posted 2013-10-10 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- patients (Experimental)
  Interventions: Procedure: electroencephalograms (EEG); Procedure: electro-myography (EMG)
- healthy volunteers (Experimental)
  Interventions: Procedure: electroencephalograms (EEG); Procedure: electro-myography (EMG)

INTERVENTIONS:
Procedure: electroencephalograms (EEG)
Procedure: electro-myography (EMG)

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is characterized clinically by abnormalities of both upper motor neurons (UMN) and lower motor neurons (LMN). The presence of UMN signs is not always easy to establish. The only technique used in routine to assess the corticospinal dysfunctions is based on transcranial magnetic stimulation (TMS). However, this technique is largely dependent on LMN state and is based on artificial motor cortex activation.

The main objective of our study project is to evaluate a new method assessing functional changes in motor system in ALS patients. By using cortico-muscular and cortico-cortical coherences, it could be possible to show modifications in both cortico-muscular relationship and in cortical activity coordination which could be related to clinical state in ALS patients. We notably expect a decrease in cortico-muscular coherence in ALS patients. Furthermore, these analyses could provide new insights in motor system plasticity phenomena. We expect a partial covering of voluntary motor command by cortical areas adjacent to primary motor cortex. Lastly, the hypothesis that an increased proportion of voluntary motor control may be assumed by ipsilateral corticospinal tract could be tested by coherence analyses.

Coherence analysis might be a useful method to detect corticospinal tract dysfunctions. This method has the advantage to be painless and not to use artificial stimulations as it is used in TMS.

ELIGIBILITY:
Inclusion Criteria:

* Patient female or male, more than 18 years,
* Patien with a diagnosis of amyotrophic lateral sclerosis according to the El Escorial criteria of Brooks et al. 1994
* Patient , the beginning of the SLA date less than 12 months,
* Patient not having a familial form of ALS,
* Patient not having cancer, autoimmune disease, liver failure, severe hypertension or untreated, severe conduction disorders or uncontrolled arrhythmia
* Patient not having a chronic psychiatric disease, dementia.
* Patient with normal visual function
* Patients receiving social coverage
* Patient have read, understood and signed an informed consent after information

Exclusion Criteria:

* Patient minor
* Patient with a familial form of ALS,
* Patient associated with severe progressive disease (cancer, autoimmune disease , liver failure )
* Patient (s) with chronic mental illness, dementia ,
* Presence of atypical clinical signs such as cerebellar ataxia , extrapyramidal signs, sensory disorders , autonomic dysfunction .
* Clinical signs of chronic respiratory failure or slow and / or forced less than 70% of the theoretical value or chronic hypercapnia than 45 mmHg vital capacity .
* Patient private freedom following a judicial or administrative decision
* Patient major Trust
* Pateinte pregnant, parturient , lactating
* Patient major in legal protection ( guardianship )
* Pateinte pregnant , parturient , lactating
* Patient hospital without consent
* Patient admitted in a health or social establishment for purposes other than research

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
recording neuronal activities | 12 months
  simultaneous recording of brain activity using electrodes attached to the scalp and muscle activities of muscles of the hands with electrodes bonded to the skin.

SECONDARY OUTCOMES:
identify plasticity phenomena | 12 months
  identify plasticity phenomena used in the cortex during the disease. The question is whether a reorganization of cortical networks could preserve, temporarily, the ability of patients to perform muscle contractions which case to determine the nature of the changes induced

CONTACTS AND LOCATIONS:
Overall Officials: LOIC MONDOLONI, Study Director — Assistance Publique Hopitaux De Marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France